CLINICAL TRIAL: NCT05354518
Title: Evaluation of the Effectiveness of Teaching Method With Simulation in Gestational Diabetes Mellitus Management
Brief Title: Teaching Method With Simulation in Gestational Diabetes Mellitus Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Esra Yılmaz, principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: sbu_yılmaz38
Record Dates: First submitted 2022-04-17; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Diabetes, Gestational
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- gestational diabetes management simulation (Experimental)
  Interventions: Behavioral: gestational diabetes management of midwifery students
- no intervention will be made (No Intervention)

INTERVENTIONS:
Behavioral: gestational diabetes management of midwifery students — Gestational diabetes management of midwifery students with a simulator
  Arms: gestational diabetes management simulation

SUMMARY:
Gestational Diabetes Mellitus is one of the common risk factors of pregnancy and occurs for the first time during pregnancy. It adversely affects maternal and fetal health and causes an increase in morbidity and mortality rates. In this context, it is very important to identify possible risks for GDM, plan, implement and evaluate initiatives, provide emergency crisis management in a short time without damage, and increase the self-confidence of midwives. In recent years, interest in simulation methods and skill acquisition training in midwifery education has increased. Research; In the management of GDM, to increase the satisfaction and self-confidence level of midwifery students in learning, to evaluate the simulation design and educational effectiveness, it was planned to use the scenario-based near-realistic simulation method in the form of randomized control-intervention quantitatively, and in qualitative design to evaluate the students' views on the method and educational effectiveness. The research will make it easier for midwifery students to intervene with the patient in a shorter time, with confidence and with sufficient clinical skills, and patient safety will be increased. In addition, it will allow the reduction of erroneous clinical practices and malpractices. This study aims to evaluate the satisfaction and self-confidence status of midwifery students and the educational effectiveness of the scenario-based simulation method with high closeness to reality in GDM management and to examine the opinions about this method to fill the gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* Being a midwifery 3rd year student and taking the "risky pregnancy" course,
* Those who have no previous clinical experience in GDM (Health College, Health Vocational High School Graduate, etc.)

Exclusion Criteria:

* To fill in the data collection forms of the study incompletely,
* Not participating in all applications of simulation training with high proximity to reality,
* Desire to leave the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-04-19 (Estimated); Primary Completion 2022-04-19 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
information evaluation form | immediately before simulation
  The information evaluation form is in a multiple-choice format consisting of 25 questions by scanning the literature by the researchers. Each question is worth 4 points.
information evaluation form | 7 weeks after the first simulation application
  The information evaluation form is in a multiple-choice format consisting of 25 questions by scanning the literature by the researchers. Each question is worth 4 points.
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the first simulation application
  The scale is a 13-item measurement tool designed to measure student satisfaction with simulation and self-confidence during practices. It is a 5-point Likert type and is scored as strongly disagree 1, disagree 2, undecided 3, agree 4, strongly agree 5.
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the second simulation application
  The scale is a 13-item measurement tool designed to measure student satisfaction with simulation and self-confidence during practices. It is a 5-point Likert type and is scored as strongly disagree 1, disagree 2, undecided 3, agree 4, strongly agree 5.
Student Satisfaction and Self-Confidence Scale in Learning | immediately after the third simulation application
  The scale is a 13-item measurement tool designed to measure student satisfaction with simulation and self-confidence during practices. It is a 5-point Likert type and is scored as strongly disagree 1, disagree 2, undecided 3, agree 4, strongly agree 5.
Simulation Design Scale | immediately after the first simulation application
  The simulation method applied and designed to the intervention group is used in the evaluation of the participants. The simulation design scale consists of 20 items in total. Evaluation of the scale is done in two stages. In the first stage, in order to evaluate whether the items used in the simulation method were given in the best way for the participant, they were expressed as strongly disagree, disagree, undecided, agree, strongly agree. In the second stage, there are statements that will determine the level of importance of the scale items for the participant, not important, partially important, undecided, important, very important. In the evaluation phase, the scale score is calculated by dividing the total and the total of the sub-dimensions by the number of items.
Simulation Design Scale | immediately after the second simulation application
  The simulation method applied and designed to the intervention group is used in the evaluation of the participants. The simulation design scale consists of 20 items in total. Evaluation of the scale is done in two stages. In the first stage, in order to evaluate whether the items used in the simulation method were given in the best way for the participant, they were expressed as strongly disagree, disagree, undecided, agree, strongly agree. In the second stage, there are statements that will determine the level of importance of the scale items for the participant, not important, partially important, undecided, important, very important. In the evaluation phase, the scale score is calculated by dividing the total and the total of the sub-dimensions by the number of items.
Simulation Design Scale | immediately after the third simulation application
  The simulation method applied and designed to the intervention group is used in the evaluation of the participants. The simulation design scale consists of 20 items in total. Evaluation of the scale is done in two stages. In the first stage, in order to evaluate whether the items used in the simulation method were given in the best way for the participant, they were expressed as strongly disagree, disagree, undecided, agree, strongly agree. In the second stage, there are statements that will determine the level of importance of the scale items for the participant, not important, partially important, undecided, important, very important. In the evaluation phase, the scale score is calculated by dividing the total and the total of the sub-dimensions by the number of items.

SECONDARY OUTCOMES:
Semi-Structured Focus Group Training Activity Evaluation Form | 7 weeks after starting the study
  It is a form consisting of 5 semi-structured questions created by the researchers after a comprehensive literature search in order to evaluate the simulation training effectiveness. With these questions, it was aimed to determine the strengths and weaknesses of training with the simulation method regarding GDM management, the opportunities/opportunities it provides and the threats and dangers created by this method.

IPD SHARING:
Plan to Share IPD: Undecided